CLINICAL TRIAL: NCT05084417
Title: ClinPRO-DERM: A Prospective, Observational Study of Clinician and Patient-reported Outcomes in Patients With Dermatological Conditions
Brief Title: A Prospective, Observational Study of Clinician and Patient-reported Outcomes in Patients With Dermatological Conditions
Acronym: ClinPRO-DERM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: OM1, Inc. (Industry)
Collaborators: American Academy of Dermatology (Unknown)
Responsible Party: Sponsor
Other Study IDs: OM1-DERM-001
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis; Dermatology; Vitiligo; Alopecia Areata; Hidradenitis Suppurativa; Psoriasis
Keywords: Registry; Patient Outcomes; Dermatological Conditions
MeSH Terms: conditions — Dermatitis, Atopic; Vitiligo; Alopecia Areata; Hidradenitis Suppurativa; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1: Alopecia Areata: Cohort 1 is limited to patients clinically diagnosed with Alopecia Areata. Patients in this cohort will receive the universal ClinROs and PROs (i.e. not disease specific) as well as additional AA-specific measures throughout the length of the study.
  Interventions: Other: N/A This is an observational study
- Cohort 2: Atopic Dermatitis: Cohort 2 is comprised of patients that have been clinically diagnosed with Atopic Dermatitis. Patients in this cohort will receive the universal PROs and ClinROs, but will also receive additional AD-specific measures throughout the length of the study.
  Interventions: Other: N/A This is an observational study
- Cohort 3: Hidradenitis Suppurativa: Cohort 3 is limited to patients clinically diagnosed with Hidradenitis Suppurativa. Patients in this cohort will receive the universal ClinROs and PROs (i.e. not disease specific) as well as additional HS-specific measures throughout the length of the study.
  Interventions: Other: N/A This is an observational study
- Cohort 4: Psoriasis: Cohort 4 is limited to patients clinically diagnosed with Psoriasis. Patients in this cohort will receive the universal ClinROs and PROs (i.e. not disease specific) as well as additional PsO-specific measures throughout the length of the study.
  Interventions: Other: N/A This is an observational study
- Cohort 5: Vitiligo: Cohort 5 is limited to patients clinically diagnosed with Vitiligo. Patients in this cohort will receive the universal ClinROs and PROs (i.e. not disease specific) as well as additional VL-specific measures throughout the length of the study.
  Interventions: Other: N/A This is an observational study

INTERVENTIONS:
Other: N/A This is an observational study — As this is an observational study, there are no interventions assigned to either cohort.

SUMMARY:
The primary goal of the study is to collect standardized patient and clinician reported outcome measures for patients diagnosed with a range of dermatological conditions in an academic clinical practice setting. By regularly measuring outcomes longitudinally in patients treated in a real-world setting, this study will provide valuable and necessary information as to the impact of both the disease and its treatments on patients over time and will inform the optimal clinical management of patients with living with dermatological disease.

DETAILED DESCRIPTION:
The study is a multi-center, longitudinal, observational study to describe longitudinal trajectories of Clinician-Reported Outcomes (ClinROs) and Patient-Reported Outcomes (PROs) in patients with select dermatological conditions. This study will collect data using validated clinical instruments and patient-reported data on the disease course of alopecia areata (AA), atopic dermatitis (AD), hidradenitis suppurativa (HS), psoriasis (PsO), and vitiligo (VL), including symptom assessments and quality of life (QoL) measures from a patient perspective, to supplement routine clinical data collected from their healthcare providers. ClinRO data will be collected at baseline and routine follow-up visits for up to two years. PRO data will be collected directly from patients at baseline and at pre-specified follow-up time points (as defined in Tables 1 - 2e) for up to two years.

The objectives of this study are:

* To describe longitudinal changes in disease activity, symptom control and both physical and mental HrQoL based on both ClinROs and PROs
* To identify patient, disease and treatment factors associated with changes in PROs over time
* To describe the association between PROs, ClinROs and clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult (defined as the age of majority in their state of residence or older) at enrollment
* Able to read and communicate in English
* Have a smart phone or other internet enabled device capable of PRO data collection
* Diagnosed with a qualifying, clinically confirmed, diagnosis of a study condition in the judgement of the treating physician at presentation
* Willing and able to provide informed consent
* Willing to participate in the collection of patient-reported outcomes for up to two years

Exclusion Criteria:

* Current (or planned) participation in an interventional clinical trial where treatment and/or management of any of the study conditions is being dictated by a protocol.
* Patient is not expected to be actively followed (i.e., seen at least annually as part of routine care) at the site for the duration of the follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (defined as at least the age of majority in their state or older) who have received a clinical diagnosis of alopecia areata, atopic dermatitis, hidradenitis suppurativa, psoriasis, or vitiligo.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Overall body surface area involvement (%BSA-AD, single score, scored 0-100) | Baseline to 2 years
  A simple measure of percent body surface area involved that complements the IGA in providing a relatively quick accurate representation of disease extent and severity.
Investigator Global Assessment (IGA, scored 0-4; clear, almost clear, mild, moderate, and severe). | Baseline to 2 years
  A 5-point IGA scale including morphologic descriptions, ranging from 0 (clear) to 4 (severe).
Dermatology Life Quality Index (DLQI, 10 items, scored 0-30) | Baseline to 2 years
  The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week
Work Productivity and Activity Impairment questionnaire (WPAI,-GH v2.0, 6 items) | Baseline to 2 years
  The questionnaire has four domains: Work Time Missed; Percent Impairment While Working; Percent Overall Work Impairment; and Percent Activity Impairment. Only one domain (Percent Activity Impairment) is completed by patients who are not currently employed
EuroQoL 5-dimension (EQ-5D; 5 items and a single VAS) | Baseline to 2 years
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Patient Health Questionnaire-2 (PHQ-2, 2 items) | Baseline to 2 years
  A simple two-item questionnaire evaluating the degree to which an individual has experienced depressed mood and anhedonia over the past two weeks. This survey is intended to screen for potential depression and is not diagnostic

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Weiss, MD, Principal Investigator — OM1, Inc.
Locations (1):
- OM1, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No